CLINICAL TRIAL: NCT01112579
Title: Determining the Feasibility of Spinal Cord Neuromodulation for the Treatment of Chronic Heart Failure
Acronym: DEFEAT-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEFEAT-HF
Record Dates: First submitted 2010-04-16; First posted 2010-04-28 (Estimated); Results first posted 2015-10-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental)
  Interventions: Device: Medtronic PrimeADVANCED Neurostimulator
- Control (Other)
  Interventions: Device: Medtronic PrimeADVANCED Neurostimulator

INTERVENTIONS:
Device: Medtronic PrimeADVANCED Neurostimulator — Heart failure therapy
  Arms: Treatment
Device: Medtronic PrimeADVANCED Neurostimulator — Medical management
  Other Names: Medical management
  Arms: Control

SUMMARY:
The purpose of this study is to determine the feasibility of spinal cord stimulation (SCS) as a chronic therapy for systolic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Left Ventricular Ejection Fraction (LVEF) of 35 percent or less
* New York Heart Association (NYHA) functional Class III at time of screening
* QRS duration less than 120 milliseconds (ms)
* Left Ventricular End Diastolic Diameter (LVEDD) of 55 millimeters (mm) to 80 mm as determined by echocardiography within the past 6 months
* Receiving stable optimal medical therapy for heart failure prior to enrollment
* Serum creatinine less than or equal to 3.0 milligrams per deciliter (mg/dL)
* 18 years of age or older
* Willing and able to comply with study procedures
* Expected lifespan greater than 12 months beyond study enrollment as assessed by physician

Exclusion Criteria:

* Interruption of thromboprophylaxis (e.g., heparin, LMWH, warfarin, aspirin, dabigatran, clopidogrel) would pose an unacceptable health risk (e.g., patient with an abnormal bleeding time), as determined by physician
* Polyneuropathy
* Requires diathermy including shortwave diathermy, microwave diathermy, or therapeutic ultrasound diathermy
* Unable to perform an exercise capacity test
* Pregnant or planning to become pregnant during this study
* Currently enrolled or plans to enroll in another investigational device or drug study that may confound the results of this study
* Had Coronary Artery Bypass Graft/Percutaneous Coronary Intervention/Bare Metal Stent (CABG/PCI/BMS) procedures within the past 90 days
* Had a heart transplant
* Has complete heart block
* Had Acute Coronary Syndrome within the past 90 days
* Has congenital heart disease with significant hemodynamic shunting
* Has chemotherapy-induced heart failure
* Has reversible cardiomyopathy
* Has severe mitral regurgitation (greater than 60 percent regurgitant fraction or greater than 0.3 centimeters squared (cm2) regurgitant orifice area)
* Has diagnosed unstable angina pectoris
* Has unstable coronary artery disease
* Has a Cardiac Resynchronization Therapy (CRT) device implanted and is receiving CRT therapy
* Has a non-Medtronic Implantable Cardioverter Defibrillator (ICD), pacemaker, or any non-transvenous defibrillation lead
* Has a Medtronic ICD whose sensing threshold cannot be programmed to 0.3mV or greater
* Has an existing neurostimulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2010-04; Primary Completion 2014-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas P Zipes, M.D., Principal Investigator — Krannert Institute of Cardiology; Heinz Theres, M.D., Principal Investigator — Charite Universitatsmedizin Berlin - Campus Charite Mitte
Locations (19):
- United States (6):
  - Miami, Florida
  - Indianapolis, Indiana
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Burlington, Vermont
  - Spokane, Washington
- Canada (2):
  - Vancouver, British Columbia
  - Victoria, British Columbia
- Prague, Czechia
- Germany (2):
  - Berlin
  - Herne
- Rome, Italy
- Netherlands (3):
  - Groningen
  - Maastricht
  - Zwolle
- South Africa (2):
  - Cape Town
  - Johannesburg
- Sweden (2):
  - Gothenburg
  - Stockholm

REFERENCES:
- [Derived] Zipes DP, Neuzil P, Theres H, Caraway D, Mann DL, Mannheimer C, Van Buren P, Linde C, Linderoth B, Kueffer F, Sarazin SA, DeJongste MJL; DEFEAT-HF Trial Investigators. Determining the Feasibility of Spinal Cord Neuromodulation for the Treatment of Chronic Systolic Heart Failure: The DEFEAT-HF Study. JACC Heart Fail. 2016 Feb;4(2):129-136. doi: 10.1016/j.jchf.2015.10.006. Epub 2015 Dec 9. PMID 26682789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 42 | 24
Completed | 41 | 21
Not Completed | 1 | 3
Not completed — Missed Visit | 1 | 1
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 42 | 24 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11) | 66 (11) | 61 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 14
  Male | 32 | 20 | 52
Region of Enrollment [Number; unit: Randomized participants]
  Canada | 3 | 0 | 3
  Czech Republic | 12 | 10 | 22
  Netherlands | 9 | 5 | 14
  Sweden | 4 | 5 | 9
  United States | 9 | 3 | 12
  Italy | 3 | 0 | 3
  South Africa | 1 | 1 | 2
  Germany | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Reduction in Left-ventricular End Systolic Volume Index (LVESVi) After 6 Months of Spinal Cord Stimulation (SCS) Therapy in the Treatment Arm Compared to the Control Arm.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Treatment | Control
Number analyzed (Participants) | 40 | 20
mL/m2 | 2.8 (16.0) | -3.6 (14.9)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.3, ANCOVA; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [-2.0 to 14.9]

2. Secondary Outcome: Characterize the Change in proBNP Between the Treatment Arm and Control Arm Through 6 Months
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment | Control
Number analyzed (Participants) | 34 | 21
pg/mL | -32.4 (994.0) | 73.8 (1468.0)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.79, ANCOVA; Mean Difference (Final Values) = -106.1, 95% CI 2-sided [-845.8 to 633.6]

3. Secondary Outcome: Characterize the Change in Peak Oxygen Uptake Between the Treatment Arm and Control Arm Through 6 Months
Time Frame: Baseline and 6 Months
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Treatment | Control
Number analyzed (Participants) | 28 | 13
mL/kg/min | 0.6 (4.1) | -0.2 (3.3)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority or Other; p = 0.93, ANCOVA; Mean Difference (Final Values) = 0.8, 95% CI 2-sided [-1.6 to 3.2]

ADVERSE EVENTS:
Arm/Group | Treatment | Control
Serious Adverse Events (participants affected / at risk) | 30/42 | 16/24
Other Adverse Events (participants affected / at risk) | 19/42 | 12/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=42) | Control (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Perforation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 2 (2)
Decompensated Heart Failure (Cardiac disorders) | 16 (33) | 7 (15)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic Cyst (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2)
Adverse Drug Reaction (General disorders) | 0 (0) | 1 (1)
Arterial Restenosis (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 2 (2) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Device Extrusion (General disorders) | 0 (0) | 1 (1)
Device Inappropriate Shock Delivery (General disorders) | 1 (1) | 0 (0)
Device Lead Damage (General disorders) | 1 (1) | 1 (1)
Lead Dislodgement (General disorders) | 3 (3) | 0 (0)
Sudden Cardiac Death (General disorders) | 2 (2) | 0 (0)
Sudden Death (General disorders) | 0 (0) | 1 (1)
Ischaemic Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium Difficile Colitis (Infections and infestations) | 0 (0) | 1 (3)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Pericarditis Infective (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (6) | 3 (3)
Pyleonephritis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gallbladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectosigmoid Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of Consiousness (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Failure Chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Endometrial Atrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry Gangrene (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic Dissection (Vascular disorders) | 1 (1) | 0 (0)
Circulatory Collapse (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=42) | Control (N=24)
Decompensated Heart Failure (Cardiac disorders) | 8 (12) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Adverse Drug Reaction (General disorders) | 2 (2) | 2 (2)
Device Stimulation Issue (General disorders) | 5 (6) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4)
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No